CLINICAL TRIAL: NCT05155748
Title: Deprescribing Inappropriate Medication in Residents Suffering From Severe Dementia: OptimaMed Long Term Care, a Demonstration Project
Brief Title: Deprescribing Intervention Among Nursing Home Residents With Major Neurocognitive Disorders
Acronym: OptimaMedLTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dre Edeltraut Kröger (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Sponsor-Investigator, Dre Edeltraut Kröger, adjunct professor, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OptimaMed-2
Record Dates: First submitted 2018-12-21; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Nursing staff, physicians and pharmacists will be invited to a continuous education - knowledge exchange session to inform them on the study rationale and the means of medication optimization.
  Pharmacists will be asked to perform medication reviews, guided by the information and tools provided, for the participating residents.
  Pharmacists' recommendations will be discussed during meetings with physician and nurses.
  Interventions: Other: Continuous education and knowledge exchange
- Control (No Intervention): Care as usual.

INTERVENTIONS:
Other: Continuous education and knowledge exchange — The intervention is educational and directed at the complete nursing home care team.
  Arms: Intervention

SUMMARY:
Canadians with neurocognitive disorders often are admitted to nursing homes when their disease reaches an advanced stage. At the end of their life, they may encounter adverse symptoms related to medications they no longer need, while they should receive comfort care. This study proposes an intervention to reduce the use of inappropriate medications among residents of nursing homes with major neurocognitive disorders. For that purpose, nursing homes' nursing staff, physicians and pharmacists will receive education and tools for the review, adjustment or discontinuation of the medications that have become inappropriate for the residents. The residents' families will receive information regarding the complexity of drug treatment for elderly patients with major neurocognitive disorders and they will be kept informed about the proposed changes to their relative's medication. The intervention is expected to reduce the medication load while improving or maintaining the residents' well-being.

DETAILED DESCRIPTION:
A quasi-experimental, cluster randomized controlled trial (CRCT) based on the results of a pilot study (). The study will take place over 6 months in 6 nursing homes (NHs) of the greater Quebec City Health Board, the Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale (CIUSSS-CN). Three NHs will be randomized to the intervention arm, three others will serve as controls, where care will be dispensed as usual. Informed consent will be sought from the representative of NH residents with major neurocognitive disorders (MNCDs).

Intervention in experimental NHs First, all members of the care teams, i.e. nursing staff, physicians and pharmacists, will receive an enriched continuous education-knowledge exchange session to inform them on the study rationale and the means of medication optimization. This session will provide tools and strategies on adjustment of certain medications (e.g. less stringent treatment goals for control of glycaemia or hypertension, alternatives to benzodiazepines). There will be an additional emphasis on tapering and discontinuation of antipsychotics. Second, the validated lists of "generally", "sometimes" or "rarely" appropriate medications for NH residents with major neurocognitive disorders (MNCDs) will be provided to the experimental NHs' staff. They will also receive algorithms on tapering of antipsychotics. The pharmacists will initiate the intervention by performing at least one medication review for each participating resident, shortly after baseline, and additional reviews if required by the participant's clinical condition. The pharmacists' medication review will result in recommendations to be discussed with nurses and the responsible physician in usual care team meetings.

Outcomes Medication regimens will be recorded over 6 months and the active medications corresponding to the lists of "generally", "sometimes" or "rarely" appropriate medications counted. At baseline and 6 months after the beginning of the intervention, participating residents will be observed for signs of discomfort (PACSLAC) and agitation (Cohen-Mansfield Agitation Inventory).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major neurocognitive disorders, OR severe dementia (stage 7 on the Reisberg Functional Assessment Staging Tool) of any type;
* Able to swallow
* Having prescribed medication

Exclusion Criteria:

- Has been at the nursing home for less than 2 months at the time of enrollment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Medication regimens between study beginning and follow-up, a compared between the intervention and the control groups. | Change from baseline to 4-6 months after patient's inclusion into study. Less medications mean a better outcome (reduction of medication load, implying deprescribing of inappropriate medications.
  List of active medications

SECONDARY OUTCOMES:
Change in level of the pain, as measured by the PACSLAC-F. | Change from baseline to six months after patient's inclusion into study.
  This is the French version of the Pain Assessment Checklist for Seniors with Limited Ability to Communicate (PACSLAC-F) observational scale for non verbal participating patients, between baseline and follow-up, as compared between the intervention and the control groups. The PACSLAC-F scale varies between 0 and 60 with 60 being the highest measure for the observation of pain expression. For the PACSLAC-F, lower scores mean better outcomes, signifying less pain.
  PACSLAC-French version (Validité et utilité clinique d'une grille d'observation (PACSLAC-F), pour évaluer la douleur chez des aînés atteints de démence vivant en milieu de soins de longue durée (1 to 60). Aubin M, Verreault R et al, Can J Aging, #1, Spring 2008
Change in level of agitation of participating patients between baseline and follow-up, as compared between the intervention and the control groups. | Change from baseline to six months after patient's inclusion into study.
  Cohen-Mansfield Agitation Inventory (CMAI) observational scale, range from 0 to 203. Lower scores mean better outcomes, signifying less discomfort.
  Cohen-Mansfield, J., Marx, M. S., & Rosenthal, A. S. (1989). A description of agitation in a nursing home. Journal of Gerontology: Medical Sciences, 44(3), M77-M84.

CONTACTS AND LOCATIONS:
Overall Officials: Edeltraut Kröger, Ph.D., Principal Investigator — CHU de Québec
Locations (1):
- Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant dat can be made available to other researchers upon personal request.

REFERENCES:
- [Background] Kroger E, Wilchesky M, Marcotte M, Voyer P, Morin M, Champoux N, Monette J, Aubin M, Durand PJ, Verreault R, Arcand M. Medication Use Among Nursing Home Residents With Severe Dementia: Identifying Categories of Appropriateness and Elements of a Successful Intervention. J Am Med Dir Assoc. 2015 Jul 1;16(7):629.e1-17. doi: 10.1016/j.jamda.2015.04.002. Epub 2015 May 13. PMID 25979776
- [Background] Wilchesky M, Mueller G, Morin M, Marcotte M, Voyer P, Aubin M, Carmichael PH, Champoux N, Monette J, Giguere A, Durand P, Verreault R, Arcand M, Kroger E. The OptimaMed intervention to reduce inappropriate medications in nursing home residents with severe dementia: results from a quasi-experimental feasibility pilot study. BMC Geriatr. 2018 Sep 4;18(1):204. doi: 10.1186/s12877-018-0895-z. PMID 30180821
- [Derived] Kroger E, Wilchesky M, Morin M, Carmichael PH, Marcotte M, Misson L, Plante J, Voyer P, Durand P. The OptimaMed intervention to reduce medication burden in nursing home residents with severe dementia: results from a pragmatic, controlled study. BMC Geriatr. 2023 Aug 28;23(1):520. doi: 10.1186/s12877-023-04222-4. PMID 37641020
- See also: Publication of the pilot study — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-018-0895-z